CLINICAL TRIAL: NCT03877055
Title: Phase I/II Clinical Trial of Copanlisib and Ibrutinib in Mantle Cell Lymphoma
Brief Title: A Study of Copanlisib and Ibrutinib in Mantle Cell Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 18-450
Record Dates: First submitted 2019-03-14; First posted 2019-03-15 (Actual); Results first posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-10

CONDITIONS: Mantle Cell Lymphoma (MCL)
Keywords: Copanlisib; Ibrutinib; 18-450
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — copanlisib; ibrutinib

STUDY DESIGN:
Intervention Model Description: This is a two stage protocol comprised of a single institution phase I dose escalation trial using standard 3+3 design and a phase II two stage Simon mini-max clinical trial.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Copanlisib and Ibrutinib (Experimental): Copanlisib is given intravenously on days 1, 8, and 15 of 28 day cycles. Ibrutinib is given orally every day on 28 days cycles. The maximum duration of treatment is 36 cycles not exceeding 36 months. In the phase II study, the cohort will expand and accrue patients at the recommended phase II dose of copanlisib and ibrutinib determined during phase I dose escalation. In a simon two stage mini-max design, an initial 18 patients will be enrolled, inclusive of 6 patients treated at MTD or RP2D from phase I study, in first stage.
  Interventions: Drug: Copanlisib; Drug: Ibrutinib

INTERVENTIONS:
Drug: Copanlisib — Treatment will be with intravenous copanlisib on days 1, 8, 15 of 28 day cycles.
Drug: Ibrutinib — Oral ibrutinib daily in 28 day cycles. A cycle is defined as 28 days of therapy.

SUMMARY:
The purpose of this study is to test the safety and any good and bad side effects of combining 2 study drugs, copanlisib and ibrutinib. This combination of drugs could shrink your Mantle Cell Lymphoma (MCL), but it could also cause side effects. Both these drugs have been given to people before, but this is the first time that they are being given together.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years of age at the time of signing Informed Consent
* Patient is able and willing to adhere to the study visit schedule and other protocol requirements
* Patient has histologically confirmed diagnosis of R/R mantle cell lymphoma who has received at least 1 line of therapy

  °Autologous stem cell transplant recipients must have adequate bone marrow recovery and transfusion independent
* Patients may have been previously treated with BTK or PI3K inhibitors:

  °If BTK/P13K inhibitors were part of their last treatment, patients must have had a best response of stable disease or better
* Patient has at least one measurable lesion (≥ 2 cm) according to RECIL criteria[37]
* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Patient has adequate bone marrow and organ function by:

  * Absolute neutrophil count (ANC) ≥ 1 x 10^9/L , independent of growth factor support for 14 days unless there is bone marrow involvement. For patients with bone marrow involvement, ANC ≥ 500/uL independent of growth factor support for 14 days
  * Platelets ≥100 x 10^9/L, or ≥50 x 10^9/L if bone marrow involvement and independent of transfusion support for 14 days in either situation
  * Hemoglobin (Hgb) ≥ 9.0 g/dL (no RBC transfusion within past 14 days)
  * International Normalized Ratio (INR) ≤ 1.5
  * Serum Creatinine ≤ 1.5 x upper limit of normal (ULN) or creatinine clearance ≥ 25 mL/min as determined by the Cockcroft-Gault equation or a 24 hour urine collection
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ ULN (or ≤ 3 x ULN if liver involved with disease
  * Total serum bilirubin ≤ ULN (or ≤ 1.5 x ULN if documented hepatic involvement; or total bilirubin ≤ 3 x ULN with direct bilirubin ≤ 1.5 x ULN in patients with documented Gilbert's Syndrome.
  * Lipase ≤ 1.5x ULN
  * LVEF ≥ 50%
  * Hemoglobin A1c ≤ 8.5%

Exclusion Criteria:

* Patient has a history of non-compliance to medical regimen or inability to grant consent
* Patient is concurrently using other approved or investigational antineoplastic agent with the exception of BTK or Pi3K inhibitors in patients who had these agents as the last line of treatment

  °Patient on BTK or P13K inhibitors will be continued on therapy as they transition to protocol therapy
* Patient has not recovered to Grade 1 or better (except alopecia) from related side effects of any prior antineoplastic therapy
* Patient has had major surgery or a wound that has not fully healed within 4 weeks of starting study drugs.
* Patients who have had chemotherapy or radiotherapy within 2 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 2 weeks earlier.
* Patients who have undergone an allogenic hematopoietic stem cell transplant
* Patient has active or history of central nervous system (CNS) disease or meningeal involvement.
* Patient has history of clinically significant interstitial lung disease and/or lung disease that severely impairs lung function (as judged by the investigator)
* Patient has history of stroke or intracranial hemorrhage ≤ 6 months from starting study drugs.
* Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
* Patient has clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification, Left Ventricular Ejection Fraction (LVEF) <50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO), unstable angina pectoris, symptomatic pericarditis, QTcF > 480 msec on the screening ECG (using the QTcF formula)
* Patient has a concurrent active malignancy. Malignancies treated with a curative intent with an expected life expectancy ≥ 5 years or a non-competing life expectancy risk are eligible (i.e. adequately treated basal or squamous cell carcinoma, non-melanomatous skin cancer, early stage breast cancer, treated prostate cancer or any other cancer from which the patient has been disease free for ≥ 3 years).
* Patient with known history of human immunodeficiency virus (HIV), or any uncontrolled active systemic infection.
* Patient has CMV viremia (peripheral blood CMV PCR positive), acute viral hepatitis (typically defined by elevated AST/ALT), or a history of chronic or active HBV or HCV infection. HBV infection is defined as having HBsAg and/or HBcAb positive test with concurrent detectable HBV DNA levels. HCV infection is defined as detectable HCV RNA levels.
* Patient requires treatment with a strong or moderate cytochrome P450 (CYP) 3A4 inhibitors, and inducers, and the treatment cannot be discontinued or switched to a different medication prior to starting study drug. Moderate and strong CYP modulators (inducers and inhibitors) should have a washout period of at least 5-6 half-lives before initiating ibrutinib or copanlisib.
* Patients with known bleeding diathesis (e.g. von Willebrand 's disease) or hemophilia
* Patient is currently receiving warfarin or other Vitamin K antagonist. Therapy with heparin, low molecular weight heparin (LMWH), or fondaparinux is allowed. Refer to Section 9.5 for Concomitant medication
* Patients with Child Pugh Class B or C hepatic cirrhosis
* Patients with any life threatening illness, medical condition or organ system dysfunction that in the opinion of the investigator could compromise the subject's safety, interfere with absorption of metabolism of study drugs or put the study outcomes at undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Connie Batlevi, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.
Supporting Information: SAP, ICF

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Copanlisib 45 mg; Ibrutinib 560 mg
- Cohort 2: Copanlisib 60 mg; Ibrutinib 560 mg
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 6 | 2
Completed | 6 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 6 | 2 | 8
Age, Continuous [Median (Full Range); unit: years] | 65 [61 to 76] | 72 [70 to 74] | 67 [61 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 5 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 2 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 2 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Complete Response
Description: using the RECIL criteria
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 6 | 2
Participants
  Complete Response | 3 | 1
  Partial Response | 2 | 1
  No Response | 1 | 0

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 5/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/2
Other Adverse Events (participants affected / at risk) | 6/6 | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=6) | Cohort 2 (N=2)
Diarrhea (Gastrointestinal disorders) | 4 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 2
Platelet count decreased (Investigations) | 4 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1
Anorexia (Metabolism and nutrition disorders) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 2
Alkaline phosphatase increased (Investigations) | 2 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 1
Fatigue (General disorders) | 2 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Neutrophil count decreased (Investigations) | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 0
Belching (Gastrointestinal disorders) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Creatinine increased (Investigations) | 0 | 1
Diabetes Mellitus Type 2 (Metabolism and nutrition disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythematous rash (non-macular, non-papular) (Skin and subcutaneous tissue disorders) | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Lip infection (Infections and infestations) | 0 | 1
Lipase increased (Investigations) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Weight loss (Investigations) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abnormal EKG (Cardiac disorders) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Edema limbs (General disorders) | 1 | 0
Edema limbs- L ankle (General disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Fever (General disorders) | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Laryngopharyngeal dysesthesia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Melena (Gastrointestinal disorders) | 1 | 0
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle strain, L pectoralis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Peripheral sensory neuropathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Serum amylase increased (Investigations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 1 | 0
Tinea pedis (Infections and infestations) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0
Urinary frequency (Renal and urinary disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-08): https://cdn.clinicaltrials.gov/large-docs/55/NCT03877055/Prot_SAP_000.pdf